CLINICAL TRIAL: NCT04806659
Title: A Phase 1, Multicenter, Safety, Pharmacokinetic, and Clinical Activity Study of SH1573 Capsules in Subjects With Refractory or Relapsed Acute Myelogenous Leukemia With an IDH2 Mutation
Brief Title: A Phase 1 Study of SH1573 Capsules in Subjects With Refractory or Relapsed Acute Myelogenous Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Sanhome Pharmaceutical, Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHC016-I-01
Record Dates: First submitted 2021-03-16; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Acute Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SH1573 Capsules (Experimental): SH1573 capsules administered orally. Multiple doses will be administered by effiacy and safety to determine the RP2D.
  Interventions: Drug: SH1573 Capsules

INTERVENTIONS:
Drug: SH1573 Capsules — Patients from each cohort will be administered SH1573 capsules every day of 28-day treatment cycles until disease progression or unacceptable toxicities.

SUMMARY:
An open label single-arm clinical trial to evaluate the safety, tolerability, PK, PD, and preliminary efficacy of SH1573 in subjects with advanced relapsed, refractory acute myelogenous leukemia that harbor an IDH2 mutation.

DETAILED DESCRIPTION:
SH1573 is an IDH2 mutation inhibitor.

This is a phase 1, open-label, multicenter, single-arm study to evaluate safety, tolerability, PK, PD, and preliminary efficacy of SH1573 capsules in treatment of subjects with advanced relapsed, refractory acute myeloid leukemias (AML) that harbor an IDH2 mutation.

The study consists of 2 parts: a dose-escalation part (Phase Ia) and a dose-expansion part (Phase Ib). The dose-escalation part will determine the MTD/R2PD. The dose-expansion part will administer the MTD/RP2D to subjects with mIDH2-positive AML.

ELIGIBILITY:
Inclusion Criteria:

* 1.Subjects aged ≥18 years.
* 2.Refractory or relapsed AML, or Untreated AML with age ≥70 years if not candidates for standard therapy.
* 3.Subjects must have documented IDH2 mutaion by central testing.
* 4.ECOG performance score of 0 to 2.
* 5.Platelet count ≥ 20,000/μL (transfusions allowed) unless due to underlying malignancy.
* 6.AST, ALT ≤ 3.0 x ULN unless due to underlying malignancy, and Serum total bilirubin ≤ 1.5 x ULN unless due to Gilbert's disease, a gene mutation in UGT1A1, or leukemic organ involvement; Serum creatinine ≤1.5 x ULN or creatinine clearance > 40 mL/min based on the Cockroft-Gault formula.
* 7.Female subjects with reproductive potential must have a negative serum pregnancy test within 72 hours prior to the start of therapy. Females of child-bearing potential and male patients should be willing to use barrier contraception during the study and until 6 months after completion of studyusing adequate contraceptive measures throughout the study.
* 8.Never participate in other clinical trial in 1 month.
* 9.Patients must sign and date written informed consent prior to admission to the study.

Exclusion Criteria:

* 1.Acute promyelocytic leukemia (APL).
* 2.Secondary AML followed by chronic myeloid leukemia (CML).
* 3.Subjects who previously received IDH2 mutation inhibitor.
* 4. Subjects who received systemic anticancer therapy or radiotherapy <14 days prior to their first day of study drug administration. (Hydroxyurea is allowed for the control of peripheral leukemic blasts)
* 5.Subjects who received an non-cytotoxic targeted drug <14 days or 5 half-lives prior to their first day of study drug administration.
* 6.Subjects who have undergone hematopoietic stem cell transplant (HSCT) within 60 days of the first dose,or subjects on immunosuppressive therapy post HSCT at the time of screening, or with clinically significant graft-versus-host disease (GVHD).
* 7.Subjects with any clinically relevant toxic effects of any prior treatment of cancer. (Subjects with residual Grade 1 toxicity are allowed with approval of the Medical Monitor.)
* 8.Subjects with clinical symptoms suggesting active central nervous system (CNS) leukemia or known CNS leukemia.
* 9.Subjects with uncontrolled severe infection that required anti-infective therapy.
* 10.Subjects with immediately life-threatening, severe complications of leukemia such as uncontrolled bleeding, pneumonia with hypoxia or shock, and/or disseminated intravascular coagulation.
* 11.Any of the following cardiac criteria:

  1. Active cardiac disease in 6 month before the first dose, such as New York Heart Association (NYHA) Class III or IV congestive heart failure, acute coronary syndrome or stroke.
  2. Left ventricular ejection fraction (LVEF) ≤ 40%.
  3. Mean resting corrected QT interval (QTcF) > 470(female) or 450(male) msec.
  4. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome.
  5. Subjects taking medications that are known to prolong the QT interval unless discontinue at least 5 half-lives before the first dose of study drug.
* 12. History of any other malignant tumor unless disease free survival ≥ 1 year (except clinically cured cervical carcinoma in situ, basal cells or squamous epithelial skin cancer).
* 13.Active infection with HIV, syphilis, hepatitis B or C.
* 14.Subjects with known dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally.
* 15.Subjects with uncontrolled hypertension (systolic blood pressure >180 mmHg or diastolic blood pressure > 100 mmHg) .
* 16.Subjects taking the sensitive cytochrome P450 (CYP) substrate medications that have a narrow therapeutic range are excluded from the study unless they can be transferred to other medications within ≥5 half-lives prior to dosing: paclitaxel (CYP2C8) warfarin, phenytoin (CYP2C9), S-mephenytoin (CYP2C19); Subjects taking breast cancer resistant protein (BCRP) transporter, OATP1B1 or OATP1B3 sensitive substrates should be excluded from the study unless they can be transferred to other medications within ≥ 5 half-lives prior to dosing.
* 17.Any disease or conditionins would compromise the safety of the patient or interfere with study assessments in the opinion of the Investigator.
* 18.female with breastfeeding.
* 19.History of hypersensitivity to any active or inactive ingredient of SH1573.
* 20.Subjects with any other conditions deemed by the Investigator to be likely to interfere with a subject's ability to sign informed consent, cooperate, or participate in the study participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2020-08-04 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Up to 28 days after first dose of study drug
  DLT is defined as an adverse event (AE) that meets protocol defined DLT criteria during cycle 1 （28 days every cycle）and is at least possibly related to study drug.
Number of Participants With Adverse Events (AEs) | From the first dose of the study drug to 30 days after the last dose of study drug
  The intensity of each AE was graded from 1 to 5 according to the NCI CTCAE Version 5.0.
Rate of CR/CRh (complete remission with incomplete hematologic recovery) | From the first dose of study drug to the time of progressive disease, assessed up to 36 months
  CR was defined as < 5% blasts in the bone marrow and full recovery of peripheral blood counts (platelets > 100 x 10^9/L and ANC > 1.0 x 10^9/L); CRh was defined as < 5% blasts in the bone marrow and partial recovery ofperipheral blood counts (platelets > 50 x 10^9/L and ANC > 0.5 x 10^9/L).

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | From the first dose of study drug to the time of progressive disease, assessed up to 36 months.
  ORR is defined as the percentage of participants achieving an overall response of CR, CRi, CRp, PR, or MLFS based on the 2003 revised IWG criteria for AML.
Complete Response (CR) Rate | From the first dose of study drug to the time of progressive disease, assessed up to 36 months
  CR was defined as < 5% blasts in the bone marrow and full recovery of peripheral blood counts (platelets > 100 x 10^9/L and ANC > 1.0 x 10^9/L).
Duration of Response(DOR) | From the first dose of study drug to the time of progressive disease, assessed up to 36 months
  DOR was defined as the time from the date of first documented response until the date of documented progression or death in the absence of disease progression.
Overall Survival | From the first dose of study drug to the end of study or death, assessed up to 36 months
  Overall survival was defined as the time from the date of first dose until death from any cause and was used to further assess the efficacy of SH1573.
Time to response (TTR) | From the first dose of study drug to the first response, assessed up to 36 months
  TTR is defined as the time from the date of first dose to the date of the first occurrence of response of CR, CRi, CRp, PR, or MLFS based on the 2003 revised IWG criteria for AML.
Proportion of non-blood transfusion dependent subjects | From the first dose of study drug to last dose of study drug, assessed up to 36 months
  It is defined as the proportion of subjects who do not need blood transfusion for any sequential period ≥8 weeks during the study treatment period.
Maximum serum drug concentration | 0, 1, 2, 4, 8, 12, 24, 48, 72 hours post-dose on single dose; 0 hour of cycle1 day 15; 0, 1, 2, 4, 8, 12, 24 hours post-dose on cycle 2 day 1; 0 hour of cycle 2 day 15 and cycle 3 day 1. Each cycle is 28 days.
  Blood samples will be obtained from all patients for determination of the maximum serum concentration of SH1573.
Area under the concentration-time curve (AUC) | 0, 1, 2, 4, 8, 12, 24, 48, 72 hours post-dose on single dose; 0 hour of cycle1 day 15; 0, 1, 2, 4, 8, 12, 24 hours post-dose on cycle 2 day 1; 0 hour of cycle 2 day 15 and cycle 3 day 1. Each cycle is 28 days.
  Blood samples will be obtained from all patients for determination of AUC of SH1573.
α-Hydroxyglutaric acid (2-HG) | 0, 24, 48 hours post-dose on single dose; Day1, Day15 pre-dose on cycle 1 and cycle 2; Day 1 pre-dose on cycle 3 and every 2 cycles afterwards. Each cycle is 28 days.
  Plasma 2-HG was measured using qualified LC-MS/MS in order to characterize the pharmacodynamic (PD) effects of SH1573.

CONTACTS AND LOCATIONS:
Overall Officials: Junmin Li, PhD, Principal Investigator — No.197 Ruijin Er Road, Shanghai, P.R China
Locations (2):
- China (2):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No